CLINICAL TRIAL: NCT02199522
Title: Clinical Observation of Titration Induction and Convention Induction of Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lihong Chen (Other)
Responsible Party: Sponsor-Investigator, Lihong Chen, Department of Anesthesia ,Sixth Affiliated hospital of Sun Yat-sen University, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DDMZ-1
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Propofol Overdose of Undetermined Intent

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- titration induction of propofol (Experimental): titration induction of propofol by Fresenius pump at the speed of 1 mg•kg-1•min-1
  Interventions: Procedure: titration induction to propofol
- convention induction of propofol (No Intervention): propofol 2mg•kg-1 intravenously by Fresenius pump at the speed of 250mg•min-1

INTERVENTIONS:
Procedure: titration induction to propofol — propofol intravenously by Fresenius pump at the speed of 1 mg•kg-1•min-1, and OAA/S scale of the patients was titrated to 1
  Arms: titration induction of propofol

SUMMARY:
As we know propofol is popular use in the anesthesia induction with kilogram and it always cause hypotension. So we compare haemodynamic changes and drug consumption between propofol titrated administration and traditional administration for anesthesia induction.

DETAILED DESCRIPTION:
GroupⅠreceived propofol 2 mg/kg intravenously by Fresenius pump at the speed of 250 mg/min, GroupⅡreceived propofol intravenously by Fresenius pump at the speed of 1 mg/kg/min, and observe's assessment of alertness and sedation(OAA/S) scale of the patients was titrated to 1, then changed to a maintenance dose

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists(ASA)Ⅰor Ⅱ and aged 18-60 yr, who were scheduled for general anesthesia.

Exclusion Criteria:

* Hypertension, Severe heart,pulmonary,brain，liver and renal dysfunction; excess obesity , predicted difficult intubation,hearing obstacles;. Allergic to propofol or its fat emulsion;addictive to sedative and other drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2014-07-28 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
systolic pressure diastolic pressure mean blood pressure | 15minutes
  before propofol dosage ,1 min after the propofol dosage, 3 min , 5 min
  , endotracheal intubation done immediately,1 min,3 min,5 min,7 min,9 min after endotracheal intubation

SECONDARY OUTCOMES:
total dosage of propofol using | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: san q Jin, docter, Principal Investigator — Department of Anesthesia ,Sixth Affiliated hospital of Sun Yat-sen University
Locations (1):
- Department of Anesthesia ,Sixth Affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China